CLINICAL TRIAL: NCT00712790
Title: Phase I/II Study of SIR-Spheres Plus Sorafenib as First Line Treatment in Patients With Non-Resectable Primary Hepatocellular Carcinoma
Brief Title: Study of SIR-Spheres Plus Sorafenib as 1st Line Treatment for Non-resectable Primary Hepatocellular Carcinoma (HCC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Singapore Clinical Research Institute (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government); Bayer Healthcare Pharmaceuticals, Inc./Bayer Schering Pharma (Industry); Sirtex Medical (Industry)
Responsible Party: Principal Investigator, Pierce K.H.Chow, MBBS MMed, FAMS, FRCSE, PhD | Senior Consultant Surgeon, Singapore General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NMRC - AHCC05
Record Dates: First submitted 2008-07-07; First posted 2008-07-10 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: First line treatment for Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sequential Radioembolization-Sorafenib (Experimental): Sorafenib (400 mg twice-daily) was initiated 14 days post-radioembolization with yttrium-90 (Y) resin microspheres given as a single procedure.
  Interventions: Drug: Sorafenib; Radiation: SIR-Spheres

INTERVENTIONS:
Drug: Sorafenib — Tablet, 400mg orally, twice daily
  Other Names: BAY 43-9006
Radiation: SIR-Spheres — one time treatment and capped at 3.0 Gbq
  Other Names: Yttrium-90 Microspheres

SUMMARY:
This Phase I/II trial will evaluate the safety and activity of chemo-radiotherapy comprising a regimen of Sorafenib chemotherapy plus SIR-Spheres yttrium-90 microspheres (chemo-radiotherapy, also known as "chemo-SIRT"), for first-line treatment of patients with primary hepatocellular carcinoma (HCC) in whom surgical resection is not feasible.

This study is designed as a prelude to a planned future randomised comparative study that will compare the efficacy of Sorafenib plus SIR-Spheres versus Sorafenib alone, in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable HCC with or without systemic metastases.
* Willing, able and mentally competent to provide written informed consent prior to any testing under this study protocol, including screening tests and evaluations that are not considered to be part of the subject's routine care.
* Aged 18 years or older of either gender and any race, religion or socioeconomic group.
* Unequivocal diagnosis of primary HCC (as defined above)
* HCC that is not amenable to surgical resection or immediate liver transplantation, or that is not optimally treatable with local ablative techniques such as radio-frequency ablation, consistent with the practice of the clinical trial centre.
* Measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥10 mm with spiral CT scan.
* ECOG performance status 0 - 1.
* Adequate haematological, renal and hepatic function as follows:
* Leukocytes ≥ 2,500/μL
* Absolute Neutrophil Count ≥ 1,500/μL
* Platelets ≥ 50,000/μL
* Haemoglobin > 9.5 g/dL
* Total bilirubin ≤ 2.0 mg/dL (SIR-Spheres should not be administered as a whole liver treatment if the total bilirubin is > 2X the institutional upper limit of normal).
* INR ≤ 2.0
* ALP ≤ 5 x institutional upper limit of normal
* AST / ALT ≤ 5 x institutional upper limit of normal
* Albumin ≥ 2.5 g/dL
* Creatinine ≤ 2.0 mg/dL
* The blood results must be less than 29 days old at the time of confirming patient eligibility to receive protocol treatment.
* Life expectancy of at least 3 months without any active treatment. This is defined as a patient who has OKUDA I or II inoperable HCC.
* Suitable for protocol treatment as determined by clinical assessment undertaken by the Investigator.
* Female patients must be either postmenopausal or, if premenopausal, must have a negative pregnancy test and agree to use two forms of contraception if sexually active during their study participation.
* Male patients must be surgically sterile, or if sexually active and having a pre-menopausal female partner then must be using an acceptable form of contraception.
* Hepatic arterial anatomy suitable for implantation of SIR-Spheres, as assessed by hepatic angiogram.
* Lung shunt fraction less than or equal to 20% as assessed by a Tc-99m macroaggregated albumin liver to lung breakthrough scan.

Exclusion Criteria:

* Had previous external beam radiation therapy to the liver.
* Any ascites or other clinical signs of liver failure, on physical examination.
* Abnormal synthetic and excretory liver function tests (LFTs) as determined by serum albumin (must be < 2.5 g/dL) and total bilirubin (must be > 2.0 mg/dL), respectively.
* Tumours amenable to surgical resection for cure at presentation.
* Greater than 20% lung shunting of the hepatic artery blood flow determined by Tc-99 MAA scan.
* Pre-assessment angiogram and Tc-99 MAA scan that demonstrates significant and uncorrectable activity in the stomach, pancreas or bowel.
* Been treated with Capecitabine within the previous 8 weeks, or who will be treated with Capecitabine within 8 weeks of treatment with SIR-Spheres, due to the possible risk of potentiating or causing liver dysfunction.
* Complete main portal vein thrombosis.
* Subjects who have had hepatic artery directed therapy.
* Subjects who have had prior chemotherapy or other medical agents used to treat hepatocellular carcinoma.
* Prior external hepatic radiation therapy for HCC, or any other concomitant therapy for HCC or any investigational agent planned while on this protocol.
* Subjects with inferior vena cava (IVC) tumour thrombus or invasion
* Currently receiving any other investigational agents for the treatment of their cancer.
* Any other concurrent malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for at least five years.
* Presence of clinical signs of CNS metastases due to their poor prognosis and because progressive neurologic dysfunction would confound the evaluation of neurologic and other adverse events.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection (except viral hepatitis), symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Any of the following contraindications to angiography and selective visceral catheterization:

  * Bleeding diathesis, not correctable by the standard forms of therapy.
  * Severe peripheral vascular disease that would preclude arterial catheterization.
  * Portal hypertension with hepatofugal flow as documented on baseline spiral CT scan.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to SIR-Spheres.
* Inability or unwillingness to understand or sign a written informed consent document (non English-speaking patients may use an interpreter).
* Female subjects who are pregnant or currently breastfeeding.
* For female subjects, unless postmenopausal or surgically sterile, unwillingness to practice effective contraception, as defined by the Investigator, during the study. The rhythm method is not to be used as the sole method of contraception.
* For male subjects, unwillingness to practice effective contraception (as defined by the Investigator) while taking part in this study, because the effect of the SIR-Spheres treatment on sperm or upon the development of an unborn child are unknown.
* Current enrolment in any other investigational drug or device study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-06; Primary Completion 2009-06 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Toxicity and safety | 2 years
Tumour response rate (liver ± any site). | 2 years

SECONDARY OUTCOMES:
Progression free survival at any site. | 2 years
Progression free survival in the liver. | 2 years
Survival | 2 years
Hepatic and extra-hepatic recurrence rate. | 2 years
Quality of life. | 2 years
Rate of downstaging to surgical resection or ablative therapy. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Pierce Chow, Phd, Study Chair — SGH
Locations (5):
- Yangon GI & Liver Centre, Yangon, Burma
- Selayang Hospital, Kuala Selangor, Malaysia
- Singapore (2):
  - Singapore General Hospital, Singapore
  - National Cancer Centre, Singapore
- Seoul National University Bundang Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Chow PK, Poon DY, Khin MW, Singh H, Han HS, Goh AS, Choo SP, Lai HK, Lo RH, Tay KH, Lim TG, Gandhi M, Tan SB, Soo KC; Asia-Pacific Hepatocellular Carcinoma Trials Group. Multicenter phase II study of sequential radioembolization-sorafenib therapy for inoperable hepatocellular carcinoma. PLoS One. 2014 Mar 10;9(3):e90909. doi: 10.1371/journal.pone.0090909. eCollection 2014. PMID 24614178
- See also: AHCC Trial Group — http://www.scri.edu.sg/index.php/ahcc-introduction